CLINICAL TRIAL: NCT07359391
Title: Dual Approach External Oblique Fascial Plane Block Versus Erector Spinae Plane Block for Post Operative Analgesia in Percutaneous Nephrolithotomy
Acronym: BLOCK-PCNL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amira S kenawy ,md, Lecturer of Anesthesia, Intensive Care, and Pain Management, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZU_IRB# 1985 /13-Jan-2026; ZU_IRB# 1985 /13-Jan-2026 (Other: Faculty of Medicine, Zagazig University, Egypt)
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones
Keywords: Percutaneous Nephrolithotomy; Postoperative Analgesia; Dual Approach External Oblique Fascial Plane Block; Erector Spinae Plane Block; Pain Management
MeSH Terms: conditions — Kidney Calculi; Agnosia | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and postoperative outcome assessors are blinded to group allocation. Randomization is performed using sealed opaque envelopes opened by an anesthesiologist not involved in postoperative assessment. The anesthesiologist performing the block is not blinded due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm Name: Dual External Oblique Fascial Plane Block Arm Type: Experimental (Experimental): Participants receive ultrasound-guided dual-approach (lateral and costal) external oblique fascial plane block in addition to standard general anesthesia for percutaneous nephrolithotomy.
  Interventions: Procedure: Dual External Oblique Fascial Plane Block
- Erector Spinae Plane Block (Experimental): Participants receive ultrasound-guided erector spinae plane block in addition to standard general anesthesia for percutaneous nephrolithotomy.
  Interventions: Procedure: Erector Spinae Plane Block
- General Anesthesia Only (Active Comparator): articipants receive routine general anesthesia according to institutional standard analgesic protocol without the addition of any regional anesthesia technique.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Ultrasound-guided erector spinae plane block performed with local anesthetic in addition to standard general anesthesia for percutaneous nephrolithotomy.
  Arms: Erector Spinae Plane Block
Procedure: Dual External Oblique Fascial Plane Block — Ultrasound-guided dual-approach (lateral and costal) external oblique fascial plane block performed using local anesthetic in addition to standard general anesthesia for percutaneous nephrolithotomy.
  Arms: Arm Name: Dual External Oblique Fascial Plane Block Arm Type: Experimental
Procedure: General Anesthesia — Routine general anesthesia according to institutional standard anesthetic and analgesic protocol without the addition of any regional anesthesia technique.
  Arms: General Anesthesia Only

SUMMARY:
Here is a **patient-friendly, ClinicalTrials.gov-compliant Brief Summary** written in **plain language**, avoiding technical jargon as much as possible while remaining accurate.

You can **copy-paste this directly** into the **Brief Summary** field.

* **Brief Summary**

Percutaneous nephrolithotomy (PCNL) is a common surgical procedure used to remove large kidney stones. Patients often experience moderate to severe pain after this surgery due to the surgical incision and irritation of the kidney and surrounding tissues. Effective pain control after PCNL is important to improve patient comfort, reduce the need for opioid medications, and enhance recovery.

Several regional anesthesia techniques have been developed to reduce postoperative pain. Two of these techniques are the dual-approach external oblique fascial plane block and the erector spinae plane block. Both techniques involve injecting a local anesthetic near specific muscle planes using ultrasound guidance to reduce pain signals from the surgical area. However, it is not yet clear which of these two techniques provides better pain relief after PCNL.

This study aims to compare the effectiveness of the dual-approach external oblique fascial plane block and the erector spinae plane block in controlling pain after PCNL surgery. Adult patients scheduled for PCNL will be randomly assigned to receive one of the two nerve block techniques or standard general anesthesia alone. Pain levels, additional pain medication requirements, patient satisfaction, and any block-related complications will be assessed during the first 24 hours after surgery.

The results of this study may help determine the most effective regional anesthesia technique for improving postoperative pain management in patients undergoing PCNL.

DETAILED DESCRIPTION:
Here is a **ClinicalTrials.gov-compliant Detailed Description** that is **clear, structured, non-duplicative**, and suitable for reviewers.

It expands on the Brief Summary **without repeating it**, focuses on **study design, interventions, and assessments**, and avoids excessive technical detail already covered elsewhere.

You can **copy-paste this directly** into the **Detailed Description** field.

* **Detailed Description**

This prospective, randomized, double-blind controlled clinical study is designed to compare the postoperative analgesic efficacy of two ultrasound-guided regional anesthesia techniques-the dual-approach external oblique fascial plane block and the erector spinae plane block-in adult patients undergoing percutaneous nephrolithotomy (PCNL).

Eligible patients aged 18-65 years with American Society of Anesthesiologists (ASA) physical status I or II, scheduled for unilateral PCNL under general anesthesia, will be enrolled after obtaining written informed consent. Participants will be randomly allocated in a 1:1:1 ratio into three groups: one group receiving the dual-approach external oblique fascial plane block, a second group receiving the erector spinae plane block, and a control group receiving general anesthesia alone according to the institutional standard analgesic protocol. Randomization will be performed using a computer-generated sequence, with allocation concealment ensured by sealed opaque envelopes. Outcome assessors and data analysts will be blinded to group allocation.

All patients will receive standardized general anesthesia. The regional blocks, when assigned, will be performed under ultrasound guidance using local anesthetic within safe dosage limits, following aseptic precautions. The dual-approach external oblique fascial plane block will involve injections at both the lateral abdominal wall and costal margin, while the erector spinae plane block will be performed at the thoracic paraspinal level. No regional anesthesia technique will be administered to patients in the control group.

Postoperative pain will be evaluated using the visual analog scale (VAS) at predefined time points during the first 24 hours after surgery. The primary outcome measure is postoperative pain intensity as assessed by VAS. Secondary outcome measures include total opioid (nalbuphine) consumption during the first 24 hours, intraoperative nociceptive responses as reflected by changes in heart rate and mean arterial pressure, patient satisfaction with pain management, and the incidence of block-related or anesthesia-related complications.

Rescue analgesia will be administered according to a predefined protocol when pain scores exceed the accepted threshold. All adverse events and complications related to the regional anesthesia techniques or general anesthesia will be monitored and documented throughout the intraoperative and postoperative periods.

The findings of this study are expected to clarify the relative effectiveness and safety of these two interfascial plane blocks for postoperative pain management following PCNL and may help guide clinical practice in regional anesthesia for urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) physical status I or II

Body mass index (BMI) between 18 and 35 kg/m²

Scheduled for unilateral percutaneous nephrolithotomy (PCNL)

Ability to understand the study protocol and provide written informed conse

Exclusion Criteria:Refusal to participate

Known allergy or hypersensitivity to local anesthetics

Infection at the site of block injection

Coagulopathy or bleeding disorders

Chronic pain syndrome or long-term opioid use

Severe hepatic, renal, or cardiac disease

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Intensity | First 24 hours postoperatively
  Postoperative pain will be assessed using the Visual Analog Scale (VAS; 0-10), where 0 indicates no pain and 10 indicates the worst imaginable pain, measured at predefined time points during the first 24 hours after surgery.